CLINICAL TRIAL: NCT05707130
Title: Effects of Gaze Stabilization Exercises on Dizziness, Balance and Quality of Life in Patients With Cervical Spondylosis.
Brief Title: Effects of Gaze Stabilization Exercises on Dizziness, Balance and Quality of Life in Cervical Spondylosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0218
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Dizziness; Balance; Distorted; Cervical Spondylosis
Keywords: Dizziness; Balance; Distorted; Cervical Spondylosis
MeSH Terms: conditions — Dizziness; Spondylosis

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to intervention groups by randomization. The patients in group A will be given gaze stabilization exercises and habituation exercises along with neck isometrics for 4 weeks. The patients in group B will be given neck isometrics for treatment of cervical spondylosis for 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gaze stabilization exercises group (Experimental): Experimental group will receive Vestibulo ocular reflex VOR / gaze stabilization exercise, Static neck exercise, and Habituation exercise. Neck isometric exercises like isometric flexion, extension, lateral bending will be performed.
  Interventions: Other: gaze stabilization exercises
- control group (Active Comparator): Patients in Conventional group will get neck isometric exercises like isometric flexion, extension, lateral bending.
  Interventions: Other: neck isometrics

INTERVENTIONS:
Other: gaze stabilization exercises — patients will perform gaze stabilization exercise, Static neck exercise, and Habituation exercise. Neck isometric exercises like isometric flexion, extension, lateral bending will be performed.
  Arms: gaze stabilization exercises group
Other: neck isometrics — Patients in Conventional group will get neck isometric exercises like isometric flexion, extension, lateral bending.
  Arms: control group

SUMMARY:
To determine the effects of gaze stabilization exercises on dizziness, balance and quality of life in patients with cervical spondylosis.

DETAILED DESCRIPTION:
A randomized controlled trial will be performed in which total 32 patients with cervical spondylosis will be included. The data will be collected from Riphah rehabilitation centre Lahore and Ittefaq hospital Lahore. The duration of study will be ten months. Dizziness handicap inventory, Romberg test and Vestibular Disorders Activities of Daily Living Scale will be used as data collection tools.

Data collection will be started after taking informed consent from all patients.

Patients will be allocated to intervention groups by randomization. The patients in group A will be given gaze stabilization exercises and habituation exercises along with neck isometrics for 4 weeks. The patients in group B will be given neck isometrics for treatment of cervical spondylosis for 4 weeks. After data collection, analysis of pre and post values will be done by using SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Pre diagnosed from orthopedic doctor with cervical spondylosis
* Complaining of cervicogenic dizziness confirmed with positive results to the tests namely Romberg's test, dizziness handicap inventory

Exclusion Criteria:

* Patients with cervical radiculopathy
* Any drug allergy and neurological deficits were excluded from the study.
* Dizziness due to ear infection and due to BPPV

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Romberg Test | 9 months
  The Romberg test is a test that measures your sense of balance.
Dizziness Handicap Inventory | 9 months
  The DHI contains 25 items, and a total score (0-100 points) is obtained by summing ordinal scale responses, higher scores indicating more severe handicap. The scale was developed to capture various sub-domains of self- perceived handicap and comprises 7 physical, 9 functional, and 9 emotional questions. Item scores are summed. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional) and a minimum score of 0. The higher the score, the greater the perceived handicap due to dizziness.
Vestibular Disorders Activities of Daily Living Scale | 9 months
  The scale evaluates the effects of vertigo and balance disorders on independence in everyday activities of daily living. The tool is designed to be useful for evaluating functional limitation and perceived handicap and disability before and after therapeutic intervention. The scale evaluates the effects of vertigo and balance disorders on independence in everyday activities of daily living. The scale 28- item self-report questionnaire that is broken down into 3 subscales:
  1. Functional- evaluates the individual's perception of basic self-maintenance tasks
  2. Ambulatory-evaluates perception of mobility related tasks
  3. Instrumental-evaluates self-perception in higher-level, more socially complex tasks

CONTACTS AND LOCATIONS:
Overall Officials: Zeest Hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun Y, Muheremu A, Tian W. Atypical symptoms in patients with cervical spondylosis: Comparison of the treatment effect of different surgical approaches. Medicine (Baltimore). 2018 May;97(20):e10731. doi: 10.1097/MD.0000000000010731. PMID 29768345
- [Background] Reddy RS, Tedla JS, Dixit S, Abohashrh M. Cervical proprioception and its relationship with neck pain intensity in subjects with cervical spondylosis. BMC Musculoskelet Disord. 2019 Oct 15;20(1):447. doi: 10.1186/s12891-019-2846-z. PMID 31615495
- [Background] Meng Z, Yu J, Luo C, Liu X, Jiang W, Yu L, Huang R. Anterior Cervical Spondylosis Surgical Interventions are Associated with Improved Lordosis and Neurological Outcomes at Latest Follow up: A Meta-analysis. Sci Rep. 2017 Jun 30;7(1):4407. doi: 10.1038/s41598-017-04311-6. PMID 28667278
- [Background] Lv Y, Tian W, Chen D, Liu Y, Wang L, Duan F. The prevalence and associated factors of symptomatic cervical Spondylosis in Chinese adults: a community-based cross-sectional study. BMC Musculoskelet Disord. 2018 Sep 11;19(1):325. doi: 10.1186/s12891-018-2234-0. PMID 30205836